CLINICAL TRIAL: NCT00342589
Title: Studies of Human Pneumocystis Infection
Brief Title: New Techniques for Using a Saline Wash as a Diagnostic Tool for Pneumocystis Pneumonia
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 990084; 99-I-0084
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-12-30

CONDITIONS: Pneumocystis Infection; Infection; Pneumonia, Pneumocystis; Lung Disease, Fungal; Mycoses
Keywords: Pneumocystis; HIV; Oral Wash; PCR; Drug Resistance; Natural History
MeSH Terms: conditions — Pneumocystis Infections; Infections; Pneumonia, Pneumocystis; Lung Diseases, Fungal; Mycoses

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Volunteers: Individuals exposed to environmental or person-to-person sources of organisms, including healthy volunteers, health care professionals, patient families, or other patients in health care facilities
- Patients: Patients immunosuppressed with acute pneumonia and are undergoing or have undergone a clinically indicated procedure to obtain a respiratory sample for diagnostic purposes.

SUMMARY:
This study will examine the effectiveness of a new laboratory method for detecting pneumocystis organisms in a salt-water (saline) oral wash. Pneumocystis infection in people with weakened immunity especially patients with HIV infection or cancer, organ transplant recipients and people receiving immune suppressing therapy can cause life-threatening pneumonia. Currently, pneumocystis infection is diagnosed by sputum analysis or bronchoalveolar lavage. For the sputum analysis, patients are induced to produce a sputum sample (liquid discharge from the lung) using a saline mist; however, many hospitals lack the expertise to perform this procedure. The second method, bronchoalveolar lavage, involves inserting a flexible tube into the lung and injecting saline to produce a specimen for diagnosis. This method, however, is time-consuming and can be uncomfortable. New techniques may allow the use of an oral wash to diagnose pneumocystis, even though an oral sample contains far fewer organisms than are obtained with the current methods. This study will examine whether new techniques, such as nucleic acid amplification, may enable a simple oral wash to be used effectively for diagnosis of pneumocystis infection.

Patients 3 years of age and older with weakened immunity who have acute pneumonia may be eligible for this study. In addition, people at increased risk of infection with pneumocystis, including health care professionals, family members of patients, and other patients in health care facilities, may participate.

Participants will have a medical history and review of medical records to determine their health status and determine if they have had recent respiratory problems or documented PCP. They will then provide an oral wash sample. For this procedure, subjects first rinse their mouth well. Then, they vigorously swish 50 milliliters of saline for 5 to 10 seconds and immediately repeat the procedure to provide two specimens. Washes may be requested daily, weekly, monthly, or for a period of time to be specified. Participants will also have two tubes of blood drawn (total of 20 milliliters, or 4 teaspoons) to test for evidence of pneumocystis.

Although no other tests are required for this protocol, participants may be asked to provide optional add'l samples, as follows:

If a sputum or bronchoalveolar lavage sample is required in the course of the patient s clinical mgmt, enough material will be obtained, if possible, for research purposes as well as what is needed for routine care.

An induced sputum sample may be requested just for this protocol. For this procedure, a mask with a saline mist is placed over the face, inducing a cough that, it is hoped, will produce sputum from the lungs.

DETAILED DESCRIPTION:
This study is designed to collect respiratory secretion specimens and blood samples to facilitate studies of human Pneumocystis infection and disease, to detect genes associated with drug resistance, and to assess strain variation. This study will also contribute information about the epidemiology of Pneumocystis by assessing normal volunteers who are exposed to Pneumocystis, e.g. health professionals, and looking at strain variation among isolates from patients and, if positives are found, from healthy volunteers. This study will potentially facilitate development of techniques that can be the basis of definitive studies on diagnosis, epidemiology, and transmission of Pneumocystis.

ELIGIBILITY:
* INCLUSION CRITERIA:

Either:

A. Patients (male or female) who are immunosuppressed with acute pneumonia and are undergoing or have undergone a clinically indicated procedure, such as bronchoscopy or sputum induction, to obtain a respiratory sample for diagnostic purposes.

or

B. Patients (male or female) who are immunosuppressed with acute pneumonia or individuals likely to be exposed to environmental or person-to-person sources of organisms, including healthy volunteers (with or without respiratory disease), health care professionals, patient families, or other patients in health care facilities who are willing to provide oral washes, nasal samples or blood samples and to consider providing an induced sputum sample.

All ages greater than or equal to 3 years.

Ability of individual or guardian to give informed consent.

EXCLUSION CRITERIA:

For enrollment under category B, any individual who cannot safely provide an oral wash or nasal samples (nasopharyngeal swabs, or nasal washes) as determined by the health care provider.

Pregnancy and age are not exclusion factors.

Nasal specimens will not be collected from children.

Ages: 3 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients (male or female) who are immunosuppressed with acute pneumonia and are undergoing or have undergone a clinically indicated procedure, such as bronchoscopy or sputum induction, to obtain a respiratory sample for diagnostic purposes. AND Patients (male or female) who are immunosuppressed with acute pneumonia or individuals likely to be exposed to environmental or person-to-person sources of organisms, including healthy volunteers (with or without respiratory disease), health care professionals, patient families, or other patients in health care facilities who are willing to provide oral washes, nasal samples or blood samples and to consider providing an induced sputum sample.
Sampling Method: Non-Probability Sample
Enrollment: 1015 (Actual)
Dates: Start 1999-09-28 (Actual)

PRIMARY OUTCOMES:
Collection of Pneumocystis samples | July 2018
  Collection of Pneumocystis samples for laboratory studies

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Kovacs, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kovacs JA, Masur H. Evolving health effects of Pneumocystis: one hundred years of progress in diagnosis and treatment. JAMA. 2009 Jun 24;301(24):2578-85. doi: 10.1001/jama.2009.880. PMID 19549975
- [Background] Larsen HH, Huang L, Kovacs JA, Crothers K, Silcott VA, Morris A, Turner JR, Beard CB, Masur H, Fischer SH. A prospective, blinded study of quantitative touch-down polymerase chain reaction using oral-wash samples for diagnosis of Pneumocystis pneumonia in HIV-infected patients. J Infect Dis. 2004 May 1;189(9):1679-83. doi: 10.1086/383322. Epub 2004 Apr 16. PMID 15116305
- [Background] Larsen HH, Kovacs JA, Stock F, Vestereng VH, Lundgren B, Fischer SH, Gill VJ. Development of a rapid real-time PCR assay for quantitation of Pneumocystis carinii f. sp. carinii. J Clin Microbiol. 2002 Aug;40(8):2989-93. doi: 10.1128/JCM.40.8.2989-2993.2002. PMID 12149363
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1999-I-0084.html